CLINICAL TRIAL: NCT00762021
Title: Posterior Capsule Opacification (PCO) Evaluation of the AcrySof SN60AT Lens vs. SN60WF Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Diane Houtman, Associate Director, Surgical IOL, Clinical Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-06-26
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-11

CONDITIONS: Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SN60AT (Experimental): Implantation with the AcrySof Intraocular Lens Model SN60AT
  Interventions: Device: SN60AT
- SN60WF (Active Comparator): Implantation with the AcrySof Intraocular Lens Model SN60WF
  Interventions: Device: SN60WF

INTERVENTIONS:
Device: SN60AT — Implantation with the AcrySof Intraocular Lens Model SN60AT following cataract removal.
  Arms: SN60AT
Device: SN60WF — Implantation with the AcrySof Intraocular Lens Model SN60WF following cataract removal.
  Arms: SN60WF

SUMMARY:
To assess posterior capsule opacification (PCO) in patients implanted with either the AcrySof SN60AT lens or the AcrySof SN60WF lens.

ELIGIBILITY:
Inclusion Criteria:

* patients with bilateral senile cataracts
* Age > 50 years
* Fit for hospital follow ups
* Pupils dilating > 6mm preoperatively
* Eyes expected to see 6/12 or better postoperatively

Exclusion Criteria:

* Diabetes
* On treatment for glaucoma
* Other ocular pathology
* Previous ocular surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Uncomplicated age-related bilateral cataract with the potential to see 20/40 or better in each eye
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | SN60AT | SN60WF
Started | 52 | 52
Completed | 44 | 44
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SN60AT | SN60WF | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 40 | 40 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Posterior Capsule Opacification (PCO)
Description: Thickening and opacification of the transparent membrane on which the intraocular lens is placed assessed by taking a digital retroillumination image of each eye with a dedicated retroillumination camera system. The photographs were analyzed with POCO software to measure the percentage area of PCO in the capsulorhexis area.
Time Frame: 2 years after surgery
Population: Data for all patients completing the 24 month visit were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of PCO
Arm/Group | SN60AT | SN60WF
Number analyzed (Participants) | 40 | 40
Percentage of PCO | 11.58 (20.18) [9.53 to 31.75] | 14.04 (22.15) [11.79 to 36.19]

2. Primary Outcome: 100% LogMAR Best Corrected Visual Acuity (BCVA)
Description: Best spectacle corrected vision was recorded for each eye of the patients at above follow up visits. The Visual Acuity (VA) measurement was taken under high contrast (100%), which means that there was maximum contrast between the letters on the chart and the background.
  VA is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 24 months after surgery
Population: Data for all patients completing the 24 month visit were analyzed.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | SN60AT | SN60WF
Number analyzed (Participants) | 40 | 40
LogMAR | 0.04 (0.1) [0.00 to 0.08] | 0.07 (0.2) [-0.02 to 0.04]

3. Primary Outcome: 9% LogMAR Best Corrected Visual Acuity (BCVA)
Description: Best spectacle corrected vision was recorded for each eye of the patients at above follow up visits. The Visual Acuity (VA) measurement was taken under low contrast (9%), which means that there was low contrast between the letters on the chart and the background.
  VA is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 24 months after surgery
Population: Data for all patients completing the 24 month visit were analyzed.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | SN60AT | SN60WF
Number analyzed (Participants) | 40 | 40
LogMAR | 0.42 (0.2) [0.36 to 0.48] | 0.45 (0.2) [0.29 to 0.37]

ADVERSE EVENTS:
Arm/Group | SN60AT | SN60WF
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications relating to the study should not be made without the Sponsor's prior written consent and not prior to the completion of the study. The sponsor shall be notified in writing at least 60 days prior to submission of any intention on the part of the Investigator to publish and shall provide the sponsor an opportunity to comment on any proposed publications.